CLINICAL TRIAL: NCT02573766
Title: Neuromodulation as a Treatment for Chemotherapy-Induced Peripheral Neuropathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2015-0399; 5K01AT008485-02 (NIH); NCI-2015-01923 (Registry Identifier: NCI CTRP); CCR-14-800 (Other Grant/Funding Number: Rising Tide Foundation)
Record Dates: First submitted 2015-10-07; First posted 2015-10-12 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pain
Keywords: Neurofeedback training; EEG; electroencephalograph; Questionnaires; Surveys; Chemotherapy-Induced Peripheral Neuropathy; CIPN
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurofeedback Training (Experimental): Participants participate in sessions for a minimum of 2 treatments a week for a maximum of 10 weeks for a total of 20 sessions. Participants asked to rate their pain on a scale of 0 (no pain) to 10 (the worst pain) prior to each session of neurofeedback and again at the conclusion of the session. Participants complete assessments again at the end of treatment and 1 month (+/- 2 weeks) later. Participants undergo an EEG at baseline, during each neurofeedback session, and within 7 days of the conclusion of treatment. Seven questionnaires regarding symptoms and quality of life completed at baseline, 1 week after neurofeedback sessions, and again in one month.
  Interventions: Procedure: Neurofeedback Training; Procedure: Electroencephalogram; Behavioral: Pain Scale; Behavioral: Questionnaires
- Sham Neurofeedback Training (Sham Comparator): Participants participate in sessions for a minimum of 2 treatments a week for a maximum of 10 weeks for a total of 20 sessions. Participants asked to rate their pain on a scale of 0 (no pain) to 10 (the worst pain) prior to each session of neurofeedback and again at the conclusion of the session. Participants complete assessments again at the end of treatment and 1 month (+/- 2 weeks) later. Participants undergo an EEG at baseline, during each neurofeedback session, and within 7 days of the conclusion of treatment. Seven questionnaires regarding symptoms and quality of life completed at baseline, 1 week after neurofeedback sessions, and again in one month.
  Interventions: Procedure: Neurofeedback Training; Procedure: Electroencephalogram; Behavioral: Pain Scale; Behavioral: Questionnaires
- Standard of Care (Other): Seven questionnaires regarding symptoms and quality of life completed at baseline, at follow up, and again in one month. Participants receive EEG at baseline, 1 week after neurofeedback group completes sessions, and again in one month.
  Interventions: Procedure: Electroencephalogram; Behavioral: Questionnaires

INTERVENTIONS:
Procedure: Neurofeedback Training — Neurofeedback Group + Sham Neurofeedback Group: Participants participate in sessions for a minimum of 2 treatments a week for a maximum of 10 weeks for a total of 20 sessions.
  Arms: Neurofeedback Training; Sham Neurofeedback Training
Procedure: Electroencephalogram — Participants undergo an EEG at baseline, during each neurofeedback session, within 7 days of the conclusion of treatment, and again in one month.
  Standard of care group receives EEG at baseline, 1 week after neurofeedback group completes sessions, and again in one month.
  Other Names: EEG
Behavioral: Pain Scale — Participants in neurofeedback groups asked to rate their pain on a scale of 0 (no pain) to 10 (the worst pain) prior to each session of neurofeedback, and again at the conclusion of the session.
  Other Names: Questionnaire; Survey
  Arms: Neurofeedback Training; Sham Neurofeedback Training
Behavioral: Questionnaires — Seven questionnaires regarding symptoms and quality of life completed at baseline, 1 week after neurofeedback sessions, and again in one month.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if using a type of non-invasive therapy called neurofeedback training can help teach patients with peripheral neuropathy how to change their own brain waves to lower their perception of neuropathy and help improve their overall quality of life.

Neurofeedback training is a type of therapy that uses an electroencephalograph (EEG) and a computer software program to measure brain wave activity.

This is an investigational study. The equipment used for neurofeedback training is FDA approved and commercially available. Using neurofeedback equipment to teach patients ways to modify their own brain waves to lower the perception of symptoms and improve quality of life is considered investigational.

Up to 99 participants over the age of 18 will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Baseline Tests:

If you agree to take part in this study, you will have the following baseline tests:

* You will complete 7 questionnaires about your symptoms, how you have been feeling, and your general quality of life. It should take about 20 minutes to complete.
* Basic information about you (such as your age and education level) will also be collected.
* You will have an EEG to measure the electrical activity of your brain. During the EEG, researchers will place a cap containing 19 electrodes on your scalp and 1 electrode on each earlobe. The electrodes will measure and record your brain wave activity, similar to the way a doctor listens to your heart beat from the surface of your skin. The EEG should take about 45 minutes to complete.

Study Groups:

After completing the baseline tests, you will be randomly assigned (as in the roll of a dice) to 1 of 3 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If you are assigned to Group 1, you will receive traditional neurofeedback training. Traditional neurofeedback training rewards you based on your own brain's activity.
* If you are assigned to Group 2, you will receive sham neurofeedback training. Sham neurofeedback training does not use your own brainwaves. In sham neurofeedback, you will be training from the brainwaves of another person who does not have neuropathy. Sham neurofeedback is not designed to help train your brainwaves. It is designed to be compared with traditional neurofeedback to learn if traditional neurofeedback has any real effect. If you have any questions about how sham neurofeedback is designed to work, talk with the study doctor or study staff.
* If you are assigned to Group 3, you will continue to receive standard care. You will not take part in the neurofeedback training, but you will take part in the follow-up visits (described below).

If you are assigned to Groups 1 or 2, you will not be told if you are receiving traditional neurofeedback training or sham training.

Neurofeedback Training (Groups 1 and 2):

You will have at least 2 neurofeedback training sessions each week for up to 10 weeks (20 training sessions total). The training sessions may take place on any 2 days of the week and may be up to 5 times a week, if you are interested in training more quickly. The study doctor will discuss the option of training faster with you.

Each neurofeedback training session should take about 1 hour to complete.

During each session, you will have an EEG while you sit quietly, relax, and watch a computer screen. The screen will be blank at first and then a series of pictures will appear. The pictures will change as your brainwaves change. You may also be shown pictures of flowers, bridges, mountains, and so on. You may be asked to play small games, for example a Pac-Man type game in which a small character moves around a maze. You will be able to choose to either view pictures or play a game.

When researchers see that your brain waves change in the way they are looking for, you will be "rewarded." When you are rewarded you will see a pretty picture on screen and you will hear a beep.

A neurotherapist will be present during each session to make sure you do not fall asleep and that you are relaxed during the procedure.

At each neurofeedback training session, you will also be asked to rate your neuropathic symptoms on a scale of 0-10 before you begin the neurofeedback training and again after the session is complete. This should only take a few minutes.

Length of Participation:

Your active participation on this study will be over after follow-up. If you are in Groups 2 or 3, you may be able to stay on study for an additional 4 months if you agree to Optional Procedure #1 (described below).

Follow-Up (All groups):

Within 1 week after your last neurofeedback training session and again about 1 month later:

* You will fill out the same 7 questionnaires you completed at baseline.
* You will have an EEG. If you are in Group 3, you will have this EEG about 1 week after Group 1 has completed their neurofeedback training.
* After you have completed the assessment 1 month later, you will be told which group you were in and offered neurofeedback if you were in the sham group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and read English, sign a written informed consent, and be willing to follow protocol requirements.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
3. Pain score >/= 4 on a 0-10 numeric pain scale and/or grade 3 neuropathic symptoms according to the National Cancer Institute's 4 point grading scale.
4. Neuropathic symptoms must be related to chemotherapy (in the opinion of the treating physician).
5. Patients must report neuropathic pain for a minimum of 3 months.
6. No plans to change pain medication regimen during the course of the study.
7. Off active chemotherapy treatment for minimum of 6 months.
8. Willing to come to MD Anderson for the therapy sessions; or willing to participate in the therapy sessions at their homes and live within a 45 minute drive of MDA main campus; or can participate in the therapy sessions from one of MDA's Regional Care Centers.
9. Patients who are 18 years of age or above
10. Patients who have a diagnosis of breast cancer.

Exclusion Criteria:

1. Patients who are taking any antipsychotic medications.
2. Patients with active central nervous system (CNS) disease, such as clinically-evident metastases or leptomeningeal disease, dementia, or encephalopathy.
3. Patients who have ever been diagnosed with bipolar disorder or schizophrenia.
4. Patients with known, previously diagnosed peripheral neuropathy from causes other than chemotherapy.
5. Patients who have a history of head injury or who have known seizure activity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Effects of Active, Deactivated, and No Neurofeedback (NF) on Symptoms of Chemotherapy-Induced Peripheral Neuropathy (CIPN) | 4 months
  Pain Quality Assessment Scale (PQAS) used to evaluate responses in each group.

SECONDARY OUTCOMES:
Effects of Neurofeedback on the Cortical and Subcortical Regions of the Pain Matrix Associated with Chemotherapy-Induced Peripheral Neuropathy (CIPN) | 4 months
  Changes in neuromodulation assessed using a quantitative EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org